CLINICAL TRIAL: NCT01152385
Title: A 4-month Treatment, Randomized, Double-blind, Placebo-Controlled, Multi-centre, Parallel-Group Phase 2 Study to Evaluate Efficacy, Safety and Tolerability of Different Dosing Regimens of AZD1656 as Monotherapy in Japanese Type 2 Diabetes Mellitus Patients
Brief Title: Japan Dose Regimen Study of AZD1656 in Japanese Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1020C00016
Record Dates: First submitted 2010-06-10; First posted 2010-06-29 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Japanese; phase 2; AZD1656; efficacy; dose regimen; pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- high (Experimental): AZD1656 titration 40 - 80 - 140 - 200 mg (daily dose)
  Interventions: Drug: AZD1656
- Middle (Experimental): AZD1656 titration 20 - 40 - 80 - 140 mg (daily dose)
  Interventions: Drug: AZD1656
- low (Experimental): AZD1656 titration 10 - 20 - 40 - 80 mg (daily dose)
  Interventions: Drug: AZD1656
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1656 — Oral tablet administered twice daily during 4 months
  Arms: Middle; high; low
Drug: Placebo — administered twice daily during 4 months
  Arms: 4

SUMMARY:
The purpose of this study is to compare the effect on glucose control of 3 different AZD1656 dosing regimens with placebo in Japanese type 2 diabetes mellitus (T2DM) patients, as evaluated by the change in HbA1c from baseline to the end of treatment at 4 months.

ELIGIBILITY:
Inclusion Criteria:

* women of non-childbearing potential.
* Provision of informed consent prior to any study specific procedures
* Naïve T2DM patients with HbA1c ≥ 7.5% but ≤ 10% or T2DM Patients treated with one or two oral anti-hyperglycaemic agent(s) with HbA1c ≥ 7.5% but ≤ 9.5% at enrolment visit (Visit1)

Exclusion Criteria:

* Clinically relevant medical history or concurrent disease such as cardiovascular disease, renal disease, hepatic disease and haematological disease.
* The investigator(s) judged that the Subject should not participate in the study according to screening test or medical history.
* Participation in another clinical trial and/or intake of another investigational drug within the last 30 days prior to enrolment visit

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Leonsson-Zachrisson, Study Director — AstraZeneca
Locations (3):
- Japan (3):
  - Research Site, Osaka
  - Research Site, Suita
  - Research Site, Tokyo

REFERENCES:
- [Derived] Kiyosue A, Hayashi N, Komori H, Leonsson-Zachrisson M, Johnsson E. Dose-ranging study with the glucokinase activator AZD1656 as monotherapy in Japanese patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2013 Oct;15(10):923-30. doi: 10.1111/dom.12100. Epub 2013 Apr 22. PMID 23522182

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment: 224 Study Start Date: May 2010 Study Completion Date: May 2011 Primary Completion Date: May 2011 (Final data collection date for primary outcome measure)
Pre-assignment Details: Wash-out period for patients treated with anti-diabetes treatment at enrolment.
Groups:
- High Dose: 200 mg (daily dose)
- Middle Dose: 140 mg (daily dose)
- Low Dose: 80 mg (daily dose)
- Placebo: Placebo
Period: Overall Study
Arm/Group | High Dose | Middle Dose | Low Dose | Placebo
Started | 55 | 58 | 56 | 55
Completed | 46 | 52 | 51 | 50
Not Completed | 9 | 6 | 5 | 5
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Study-specific withdrawal criteria | 1 | 1 | 2 | 0
Not completed — Other | 4 | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose | Middle Dose | Low Dose | Placebo | Total
Number analyzed (Participants) | 55 | 58 | 56 | 55 | 224
Age Continuous [Mean (Standard Deviation); unit: Years] | 57 (9) | 55 (9) | 55 (10) | 57 (9) | 56 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 8 | 9 | 32
  Male | 48 | 50 | 48 | 46 | 192

OUTCOME MEASURES:

1. Primary Outcome: Change in Haemoglobin A1c (HbA1c)
Time Frame: from baseline to 4 months
Population: The analysis population was prior to rescue treatment (FAS)
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- Arm 1 - High Dose: AZD1656 titration 40 - 80 - 140 - 200 mg (daily dose)
- Arm 2 - Middle Dose: AZD1656 titration 20 - 40 - 80 - 140 mg (daily dose)
- Arm 3 - Low Dose: AZD1656 titration 10 - 20 - 40 - 80 mg (daily dose)
- Arm 4 - Placebo Dose: Placebo
Arm/Group | Arm 1 - High Dose | Arm 2 - Middle Dose | Arm 3 - Low Dose | Arm 4 - Placebo Dose
Number analyzed (Participants) | 55 | 58 | 54 | 55
Percentage | 0.0 (1.2) | -0.3 (1.3) | 0.1 (1.2) | 0.2 (0.7)

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Time Frame: from baseline to 4 months
Population: The analysis population was prior to rescue treatment (FAS)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1 - High Dose | Arm 2 - Middle Dose | Arm 3 - Low Dose | Arm 4 - Placebo Dose
Number analyzed (Participants) | 55 | 58 | 56 | 55
mg/dL | 9 (42) | 6 (45) | 1 (36) | 16 (28)

3. Secondary Outcome: Number of Responders in Terms of HbA1C ≤ 7%
Time Frame: at 4th month
Population: The analysis population was prior to rescue treatment (FAS)
Measure: Number; unit: Participants
Groups:
- Arm 1 - High: AZD1656 titration 40 - 80 - 140 - 200 mg (daily dose)
- Arm 2 - Middle: AZD1656 titration 20 - 40 - 80 - 140 mg (daily dose)
- Arm 3 - Low: AZD1656 titration 10 - 20 - 40 - 80 mg (daily dose)
- Arm 4 - Placebo: Placebo
Arm/Group | Arm 1 - High | Arm 2 - Middle | Arm 3 - Low | Arm 4 - Placebo
Number analyzed (Participants) | 55 | 58 | 54 | 55
Participants | 7 | 16 | 7 | 1

4. Secondary Outcome: Number of Responders in Terms of HbA1C ≤ 6.5%
Time Frame: at 4th month
Population: The analysis population was prior to rescue treatment (FAS)
Measure: Number; unit: Participants
Arm/Group | Arm 1 - High | Arm 2 - Middle | Arm 3 - Low | Arm 4 - Placebo
Number analyzed (Participants) | 55 | 58 | 54 | 55
Participants | 2 | 8 | 2 | 0

5. Secondary Outcome: Percentage Change in Low-density Lipoprotein Cholesterol (LDL-C)
Time Frame: from baseline to 4 months
Population: The analysis population was prior to rescue treatment (FAS)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Arm 1 - High | Arm 2 - Middle | Arm 3 - Low | Arm 4 - Placebo
Number analyzed (Participants) | 55 | 58 | 56 | 55
Percentage | 8.9 (19.9) | 7.7 (18.8) | 4.0 (15.6) | 5.8 (18.4)

6. Secondary Outcome: Percentage Change in High-density Lipoprotein Cholesterol (HDL-C)
Time Frame: from baseline to 4 months
Population: The analysis population was prior to rescue treatment (FAS)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Arm 1 - High | Arm 2 - Middle | Arm 3 - Low | Arm 4 - Placebo
Number analyzed (Participants) | 55 | 58 | 56 | 55
Percentage | 8.8 (18.0) | 8.7 (12.9) | 11.6 (12.7) | 8.5 (12.5)

7. Secondary Outcome: Percentage Change in Triglycerides
Time Frame: from baseline to 4 months
Population: The analysis population was prior to rescue treatment (FAS)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Arm 1 - High | Arm 2 - Middle | Arm 3 - Low | Arm 4 - Placebo
Number analyzed (Participants) | 55 | 58 | 56 | 55
Percentage | 10.8 (44.0) | 25.0 (58.5) | 6.7 (29.4) | 18.1 (46.8)

8. Secondary Outcome: Change in High-sensitivity C-reactive Protein (Hs-CRP)
Time Frame: from baseline to 4 months
Population: The analysis population was prior to rescue treatment (FAS)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1 - High | Arm 2 - Middle | Arm 3 - Low | Arm 4 - Placebo
Number analyzed (Participants) | 55 | 58 | 54 | 55
mg/dL | 0.058 (0.138) | 0.021 (0.117) | 0.033 (0.125) | -0.007 (0.115)

ADVERSE EVENTS:
Arm/Group | High Dose | Middle Dose | Low Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/28 | 0/23
Other Adverse Events (participants affected / at risk) | 16/55 | 19/58 | 16/56 | 16/55
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=55) | Middle Dose (N=58) | Low Dose (N=56) | Placebo (N=55)
Nasopharyngitis (Infections and infestations) | 6 | 9 | 9 | 11
Bronchitis (Infections and infestations) | 2 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 2 | 2 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 2 | 0 | 0
Blood Triglycerides Increased (Investigations) | 0 | 2 | 0 | 0
Electrocardiogram T Wave Inversion (Investigations) | 0 | 0 | 2 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Asthenopia (Eye disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No